CLINICAL TRIAL: NCT05301959
Title: Evaluation of the Efficacy of Adding Low-intensity Percutaneous Musculoskeletal Electrolysis to the Conservative Treatment of Noninsertional Achilles Tendinopathy: a Randomized Controlled Clinical Trial
Brief Title: Efficacy of Percutaneous Electrolysis in the Treatment of Achilles Tendinopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maimonides University (Other)
Responsible Party: Principal Investigator, Santiago Marcelo d'Almeida, PT SCS PhD Candidate, Research Professor, Maimonides University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5694
Record Dates: First submitted 2022-02-27; First posted 2022-03-31 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Achilles Tendinopathy
Keywords: tendinopathy; physiotherapy; percutaneous electrolysis
MeSH Terms: conditions — Tendinopathy

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, blinded, evaluator-blinded, controlled clinical trial will be conducted in parallel groups (experimental treatment vs. sham treatment), with a follow-up at 26 and 52 weeks after the first intervention. Non-probability and intentional sampling will be performed.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): A single weekly intervention of low intensity galvanic currents will be applied in an ultrasound-guided manner.
  Interventions: Device: low intensity percutaneous musculoskeletal electrolysis; Other: Silbernagel protocol
- Simulated group. (Sham Comparator): The application of a single weekly intervention of low intensity galvanic currents will be simulated in an echogenic way, with the equipment turned off.
  Interventions: Device: Sham application; Other: Silbernagel protocol

INTERVENTIONS:
Device: low intensity percutaneous musculoskeletal electrolysis — An acupuncture needle (0.30mm X 25mm) will be introduced into the device's strut. With the equipment on and with a base intensity of 120µA, the acupuncture needle is introduced in a proximal-distal and postero-anterior direction, in the area of the Achilles tendon body. The position of the needle will be checked with ultrasound and once the point to be treated is reached, the working intensity will be increased up to 600 µA. The emission will be maintained until the participant reports a pain of 60/100 in VAS. At that moment, the emission will be paused completely until the participant reports a sensation of at least 20/100 in VAS. After this period the emission will be continued at 600 µA. This cycle will continue until the emission lasts for more than 120 sec, continuously. At this point, the needle will be repositioned to repeat the emission protocol a maximum of 3 times in total.
  Other Names: percutaneous microelectrolysis
  Arms: Experimental group
Device: Sham application — A modification will be made in a second equipment, closing the circuit with a 10kΩ resistor inside the equipment, in the output strand chip. Allowing the simulation of emission without emitting current to the participant and without being able to appreciate any type of alteration in the handling of the equipment, by the operators. Therefore, the same steps will be followed as in the experimental group.
  Arms: Simulated group.
Other: Silbernagel protocol — The Silbernagel et al. protocol comprises several heel raising exercises with concentric and eccentric movements, performed on two legs and one leg. It is composed of 3 sets of 15 repetitions and that during the exercises allows pain to be present, but not being disabling. The exercises will be performed only once a day. The progression will be made by changing from standing exercises to monopodal support, moving from concentric-eccentric to purely eccentric loading, adding weight in a backpack (in steps of 5 kg when pain does not exceed 5 in the pain monitoring model) and finally using fast rebound exercises and plyometric exercises.
  Other Names: Silbernagel et al. Achilles tendinopathy protocol

SUMMARY:
Achilles tendinopathy (AT) is one of the most reported myotendinous pathologies due to overuse in the literature. In the general adult population, its incidence is 2.35 cases per 1,000 patients, with no difference between men and women. The international literature reports that up to 29% of patients fail with conservative treatment.

Within physiotherapy, new alternatives for the treatment of tendinopathies arise, applying electric currents percutaneously, which from a mechanical effect associated to the use of a needle and an electric effect by the use of galvanic currents, generate a local inflammatory response; activation of the central nervous system and analgesia.

The aim of the research is to evaluate the efficacy of adding low intensity percutaneous electrolysis to the treatment with a high load eccentric exercise program based on the protocol of Silbernagel et al. in adults with Achilles tendinopathy to improve its functionality.

A randomized, double-blind, blinded, evaluator-blinded, controlled clinical trial will be conducted in parallel groups (experimental treatment vs. sham treatment), with a follow-up at 26 and 52 weeks after the first intervention. Non-probability and intentional sampling will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Presence of symptoms in one or both Achilles tendons with a minimum duration of two months. In case the symptoms are bilateral, the intervention or placebo will only be administered and its results evaluated- in the limb with greater symptomatology. If it is not possible to differentiate which one presents greater pain, the right Achilles tendon will be chosen.
* Spontaneous pain of at least three points measured by a visual analog scale (VAS), reproducible by palpation between 2 and 6 cm above the insertion of the Achilles tendon in the calcaneal bone.
* Evidence of tendinopathy by MRI.
* Presence of post-static dyskinesia.
* Willingness to not perform additional treatments (such as footwear modifications, physical therapy, orthotics, injections, or surgery) for Achilles tendon pain during the conduct of the trial.
* Willingness to attempt to discontinue self-administration of medications (NSAIDs) for pain relief Achilles tendon(s) pain for at least 14 days prior to baseline assessment and during the course of the trial.

Exclusion Criteria:

* Presence or suspicion of pregnancy.
* Previous surgical intervention on the AT in the symptomatic leg(s)
* Total or partial rupture in the symptomatic AT
* Chronic ankle instability, in the foot with symptomatic tendon(s).
* Pathologies that can derive in pain in the region of the AT without being proper of the picture. (e.g.: osteoarthritis, impingement syndromes).
* Presence of arthritis or any metabolic or endocrine disorder (type 1 or 2 diabetes).
* Psychological disorders.
* Oncologic history.
* Treatment with quinolones or fluoroquinolones during the last two years.
* Treatment with statins for the control of hypercholesterolemia for more than two months
* Treatments within or at the periphery of the Achilles tendon, with anesthetics, corticosteroids or any other pharmacological agent during the last three months.
* Needle phobia
* Allergy to metal

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Victorian Institute of Sport Assessment - Achilles - Baseline | Baseline
  patient reported outcomes specifically designed for the assessment of pain and function in the achilles tendinopathy. It has a scale from 0 (worst) to 100 (best).
Victorian Institute of Sport Assessment - Achilles - Week 1 | one week at study entry
  patient reported outcomes specifically designed for the assessment of pain and function in the achilles tendinopathy. It has a scale from 0 (worst) to 100 (best).
Victorian Institute of Sport Assessment - Achilles - Week 2 | two week at study entry
  patient reported outcomes specifically designed for the assessment of pain and function in the achilles tendinopathy. It has a scale from 0 (worst) to 100 (best).
Victorian Institute of Sport Assessment - Achilles - Week 3 | three week at study entry
  patient reported outcomes specifically designed for the assessment of pain and function in the achilles tendinopathy. It has a scale from 0 (worst) to 100 (best).
Victorian Institute of Sport Assessment - Achilles - Week 4 | four week at study entry
  patient reported outcomes specifically designed for the assessment of pain and function in the achilles tendinopathy. It has a scale from 0 (worst) to 100 (best).
Victorian Institute of Sport Assessment - Achilles - Week 5 | five week at study entry
  patient reported outcomes specifically designed for the assessment of pain and function in the achilles tendinopathy. It has a scale from 0 (worst) to 100 (best).
Victorian Institute of Sport Assessment - Achilles - Week 6 | six week at study entry
  patient reported outcomes specifically designed for the assessment of pain and function in the achilles tendinopathy. It has a scale from 0 (worst) to 100 (best).
Victorian Institute of Sport Assessment - Achilles - Week 7 | seven week at study entry
  patient reported outcomes specifically designed for the assessment of pain and function in the achilles tendinopathy. It has a scale from 0 (worst) to 100 (best).
Victorian Institute of Sport Assessment - Achilles - Week 8 | eight week at study entry
  patient reported outcomes specifically designed for the assessment of pain and function in the achilles tendinopathy. It has a scale from 0 (worst) to 100 (best).
Victorian Institute of Sport Assessment - Achilles - Week 9 | nine week at study entry
  patient reported outcomes specifically designed for the assessment of pain and function in the achilles tendinopathy. It has a scale from 0 (worst) to 100 (best).
Victorian Institute of Sport Assessment - Achilles - Week 10 | ten week at study entry
  patient reported outcomes specifically designed for the assessment of pain and function in the achilles tendinopathy. It has a scale from 0 (worst) to 100 (best).
Victorian Institute of Sport Assessment - Achilles - Week 11 | eleven week at study entry
  patient reported outcomes specifically designed for the assessment of pain and function in the achilles tendinopathy. It has a scale from 0 (worst) to 100 (best).
Victorian Institute of Sport Assessment - Achilles - Week 12 | twelve week at study entry
  patient reported outcomes specifically designed for the assessment of pain and function in the achilles tendinopathy. It has a scale from 0 (worst) to 100 (best).
Victorian Institute of Sport Assessment - Achilles - Week 26 | twenty-six week at study entry
  patient reported outcomes specifically designed for the assessment of pain and function in the achilles tendinopathy. It has a scale from 0 (worst) to 100 (best).
Victorian Institute of Sport Assessment - Achilles - Week 52 | fifty-two week at study entry
  patient reported outcomes specifically designed for the assessment of pain and function in the achilles tendinopathy. It has a scale from 0 (worst) to 100 (best).

SECONDARY OUTCOMES:
visual analog scale - Baseline | Baseline
  The intensity of pain experienced during a sequence of three monopodal countermovement jumps with both hands on the waist will be evaluated on a graduated scale. A maximum of three jumps will be performed and the highest jump will be recorded. Immediately afterwards, participants will be asked to indicate with an "X" on a 100mm line the intensity of pain experienced in the Achilles tendon. It has a scale from 0 (no pain) to 100 (worst pain).
visual analog scale - Week 1 | one week at study entry
  The intensity of pain experienced during a sequence of three monopodal countermovement jumps with both hands on the waist will be evaluated on a graduated scale. A maximum of three jumps will be performed and the highest jump will be recorded. Immediately afterwards, participants will be asked to indicate with an "X" on a 100mm line the intensity of pain experienced in the Achilles tendon. It has a scale from 0 (no pain) to 100 (worst pain).
visual analog scale - Week 2 | Two week at study entry
  The intensity of pain experienced during a sequence of three monopodal countermovement jumps with both hands on the waist will be evaluated on a graduated scale. A maximum of three jumps will be performed and the highest jump will be recorded. Immediately afterwards, participants will be asked to indicate with an "X" on a 100mm line the intensity of pain experienced in the Achilles tendon. It has a scale from 0 (no pain) to 100 (worst pain).
visual analog scale - Week 3 | three week at study entry
  The intensity of pain experienced during a sequence of three monopodal countermovement jumps with both hands on the waist will be evaluated on a graduated scale. A maximum of three jumps will be performed and the highest jump will be recorded. Immediately afterwards, participants will be asked to indicate with an "X" on a 100mm line the intensity of pain experienced in the Achilles tendon. It has a scale from 0 (no pain) to 100 (worst pain).
visual analog scale - Week 4 | four week at study entry
  The intensity of pain experienced during a sequence of three monopodal countermovement jumps with both hands on the waist will be evaluated on a graduated scale. A maximum of three jumps will be performed and the highest jump will be recorded. Immediately afterwards, participants will be asked to indicate with an "X" on a 100mm line the intensity of pain experienced in the Achilles tendon. It has a scale from 0 (no pain) to 100 (worst pain).
visual analog scale - Week 5 | five week at study entry
  The intensity of pain experienced during a sequence of three monopodal countermovement jumps with both hands on the waist will be evaluated on a graduated scale. A maximum of three jumps will be performed and the highest jump will be recorded. Immediately afterwards, participants will be asked to indicate with an "X" on a 100mm line the intensity of pain experienced in the Achilles tendon. It has a scale from 0 (no pain) to 100 (worst pain).
visual analog scale - Week 6 | six week at study entry
  The intensity of pain experienced during a sequence of three monopodal countermovement jumps with both hands on the waist will be evaluated on a graduated scale. A maximum of three jumps will be performed and the highest jump will be recorded. Immediately afterwards, participants will be asked to indicate with an "X" on a 100mm line the intensity of pain experienced in the Achilles tendon. It has a scale from 0 (no pain) to 100 (worst pain).
visual analog scale - Week 7 | seven week at study entry
  The intensity of pain experienced during a sequence of three monopodal countermovement jumps with both hands on the waist will be evaluated on a graduated scale. A maximum of three jumps will be performed and the highest jump will be recorded. Immediately afterwards, participants will be asked to indicate with an "X" on a 100mm line the intensity of pain experienced in the Achilles tendon. It has a scale from 0 (no pain) to 100 (worst pain).
visual analog scale - Week 8 | eight week at study entry
  The intensity of pain experienced during a sequence of three monopodal countermovement jumps with both hands on the waist will be evaluated on a graduated scale. A maximum of three jumps will be performed and the highest jump will be recorded. Immediately afterwards, participants will be asked to indicate with an "X" on a 100mm line the intensity of pain experienced in the Achilles tendon. It has a scale from 0 (no pain) to 100 (worst pain).
visual analog scale - Week 9 | nine week at study entry
  The intensity of pain experienced during a sequence of three monopodal countermovement jumps with both hands on the waist will be evaluated on a graduated scale. A maximum of three jumps will be performed and the highest jump will be recorded. Immediately afterwards, participants will be asked to indicate with an "X" on a 100mm line the intensity of pain experienced in the Achilles tendon. It has a scale from 0 (no pain) to 100 (worst pain).
visual analog scale - Week 10 | ten week at study entry
  The intensity of pain experienced during a sequence of three monopodal countermovement jumps with both hands on the waist will be evaluated on a graduated scale. A maximum of three jumps will be performed and the highest jump will be recorded. Immediately afterwards, participants will be asked to indicate with an "X" on a 100mm line the intensity of pain experienced in the Achilles tendon. It has a scale from 0 (no pain) to 100 (worst pain).
visual analog scale - Week 11 | eleven week at study entry
  The intensity of pain experienced during a sequence of three monopodal countermovement jumps with both hands on the waist will be evaluated on a graduated scale. A maximum of three jumps will be performed and the highest jump will be recorded. Immediately afterwards, participants will be asked to indicate with an "X" on a 100mm line the intensity of pain experienced in the Achilles tendon. It has a scale from 0 (no pain) to 100 (worst pain).
visual analog scale - Week 12 | twelve week at study entry
  The intensity of pain experienced during a sequence of three monopodal countermovement jumps with both hands on the waist will be evaluated on a graduated scale. A maximum of three jumps will be performed and the highest jump will be recorded. Immediately afterwards, participants will be asked to indicate with an "X" on a 100mm line the intensity of pain experienced in the Achilles tendon. It has a scale from 0 (no pain) to 100 (worst pain).
visual analog scale - Week 26 | twenty-six week at study entry
  The intensity of pain experienced during a sequence of three monopodal countermovement jumps with both hands on the waist will be evaluated on a graduated scale. A maximum of three jumps will be performed and the highest jump will be recorded. Immediately afterwards, participants will be asked to indicate with an "X" on a 100mm line the intensity of pain experienced in the Achilles tendon. It has a scale from 0 (no pain) to 100 (worst pain).
visual analog scale - Week 52 | fifty-two week at study entry
  The intensity of pain experienced during a sequence of three monopodal countermovement jumps with both hands on the waist will be evaluated on a graduated scale. A maximum of three jumps will be performed and the highest jump will be recorded. Immediately afterwards, participants will be asked to indicate with an "X" on a 100mm line the intensity of pain experienced in the Achilles tendon. It has a scale from 0 (no pain) to 100 (worst pain).
The Foot and Ankle Ability Measure - Baseline | Baseline
  an evaluative instrument that assesses functional limitations for those with foot- and ankle-related disorders. it's a patient reported outcomes which allows to quantify sport activity and participation. It has a scale from 0 (worst) to 100 (best). It consists of 29 questions, divided into 2 subscales, activities of daily living and sports activities. The criterion for discharge is a value greater than or equal to 90 points.
The Foot and Ankle Ability Measure - Week 1 | one week at study entry
  an evaluative instrument that assesses functional limitations for those with foot- and ankle-related disorders. it's a patient reported outcomes which allows to quantify sport activity and participation. It has a scale from 0 (worst) to 100 (best). It consists of 29 questions, divided into 2 subscales, activities of daily living and sports activities. The criterion for discharge is a value greater than or equal to 90 points.
The Foot and Ankle Ability Measure - Week 2 | two week at study entry
  an evaluative instrument that assesses functional limitations for those with foot- and ankle-related disorders. it's a patient reported outcomes which allows to quantify sport activity and participation. It has a scale from 0 (worst) to 100 (best). It consists of 29 questions, divided into 2 subscales, activities of daily living and sports activities. The criterion for discharge is a value greater than or equal to 90 points.
The Foot and Ankle Ability Measure - Week 3 | three week at study entry
  an evaluative instrument that assesses functional limitations for those with foot- and ankle-related disorders. it's a patient reported outcomes which allows to quantify sport activity and participation. It has a scale from 0 (worst) to 100 (best). It consists of 29 questions, divided into 2 subscales, activities of daily living and sports activities. The criterion for discharge is a value greater than or equal to 90 points.
The Foot and Ankle Ability Measure - Week 4 | four week at study entry
  an evaluative instrument that assesses functional limitations for those with foot- and ankle-related disorders. it's a patient reported outcomes which allows to quantify sport activity and participation. It has a scale from 0 (worst) to 100 (best). It consists of 29 questions, divided into 2 subscales, activities of daily living and sports activities. The criterion for discharge is a value greater than or equal to 90 points.
The Foot and Ankle Ability Measure - Week 5 | five week at study entry
  an evaluative instrument that assesses functional limitations for those with foot- and ankle-related disorders. it's a patient reported outcomes which allows to quantify sport activity and participation. It has a scale from 0 (worst) to 100 (best). It consists of 29 questions, divided into 2 subscales, activities of daily living and sports activities. The criterion for discharge is a value greater than or equal to 90 points.
The Foot and Ankle Ability Measure - Week 6 | six week at study entry
  an evaluative instrument that assesses functional limitations for those with foot- and ankle-related disorders. it's a patient reported outcomes which allows to quantify sport activity and participation. It has a scale from 0 (worst) to 100 (best). It consists of 29 questions, divided into 2 subscales, activities of daily living and sports activities. The criterion for discharge is a value greater than or equal to 90 points.
The Foot and Ankle Ability Measure - Week 7 | seven week at study entry
  an evaluative instrument that assesses functional limitations for those with foot- and ankle-related disorders. it's a patient reported outcomes which allows to quantify sport activity and participation. It has a scale from 0 (worst) to 100 (best). It consists of 29 questions, divided into 2 subscales, activities of daily living and sports activities. The criterion for discharge is a value greater than or equal to 90 points.
The Foot and Ankle Ability Measure - Week 8 | eight week at study entry
  an evaluative instrument that assesses functional limitations for those with foot- and ankle-related disorders. it's a patient reported outcomes which allows to quantify sport activity and participation. It has a scale from 0 (worst) to 100 (best). It consists of 29 questions, divided into 2 subscales, activities of daily living and sports activities. The criterion for discharge is a value greater than or equal to 90 points.
The Foot and Ankle Ability Measure - Week 9 | nine week at study entry
  an evaluative instrument that assesses functional limitations for those with foot- and ankle-related disorders. it's a patient reported outcomes which allows to quantify sport activity and participation. It has a scale from 0 (worst) to 100 (best). It consists of 29 questions, divided into 2 subscales, activities of daily living and sports activities. The criterion for discharge is a value greater than or equal to 90 points.
The Foot and Ankle Ability Measure - Week 10 | ten week at study entry
  an evaluative instrument that assesses functional limitations for those with foot- and ankle-related disorders. it's a patient reported outcomes which allows to quantify sport activity and participation. It has a scale from 0 (worst) to 100 (best). It consists of 29 questions, divided into 2 subscales, activities of daily living and sports activities. The criterion for discharge is a value greater than or equal to 90 points.
The Foot and Ankle Ability Measure - Week 11 | eleven week at study entry
  an evaluative instrument that assesses functional limitations for those with foot- and ankle-related disorders. it's a patient reported outcomes which allows to quantify sport activity and participation. It has a scale from 0 (worst) to 100 (best). It consists of 29 questions, divided into 2 subscales, activities of daily living and sports activities. The criterion for discharge is a value greater than or equal to 90 points.
The Foot and Ankle Ability Measure - Week 12 | twelve week at study entry
  an evaluative instrument that assesses functional limitations for those with foot- and ankle-related disorders. it's a patient reported outcomes which allows to quantify sport activity and participation. It has a scale from 0 (worst) to 100 (best). It consists of 29 questions, divided into 2 subscales, activities of daily living and sports activities. The criterion for discharge is a value greater than or equal to 90 points.
The Foot and Ankle Ability Measure - Week 26 | twenty-six week at study entry
  an evaluative instrument that assesses functional limitations for those with foot- and ankle-related disorders. it's a patient reported outcomes which allows to quantify sport activity and participation. It has a scale from 0 (worst) to 100 (best). It consists of 29 questions, divided into 2 subscales, activities of daily living and sports activities. The criterion for discharge is a value greater than or equal to 90 points.
The Foot and Ankle Ability Measure - Week 52 | fifty-two week at study entry
  an evaluative instrument that assesses functional limitations for those with foot- and ankle-related disorders. it's a patient reported outcomes which allows to quantify sport activity and participation. It has a scale from 0 (worst) to 100 (best). It consists of 29 questions, divided into 2 subscales, activities of daily living and sports activities. The criterion for discharge is a value greater than or equal to 90 points.
ultrasound Shear Wave elastography - baseline | Baseline
  Shear Wave Elastography (SWS), which consists of a special ultrasound methodology that allows quantitative characterization of the elastic capacity of a tissue through the propagation velocity of the ultrasound wave. The Siemens Acuson S2000 system with a model 9L4 linear transducer will be used.
  The patients will be placed on a table in ventral decubitus and the ankle outside the plane of the table in neutral position. To determine the point to be scanned, the maximum perpendicular distance between the anterior and posterior limits of the tendon between 2 to 6 cm from the insertion in the calcaneus will be taken and this value will be reported in mm.
  The SWS value will be expressed in m/s. The range of SWS is 0-9 m/s. The standard SWS measurement window size shall be 1cm2 , with a region of interest of 3mm. Three measurements will be recorded in each plane (regions of interest) where homogeneous tissue is considered and the average value of the 6 measurements will be reported.
ultrasound Shear Wave elastography - Week 4 | four week at study entry
  Shear Wave Elastography (SWS), which consists of a special ultrasound methodology that allows quantitative characterization of the elastic capacity of a tissue through the propagation velocity of the ultrasound wave. The Siemens Acuson S2000 system with a model 9L4 linear transducer will be used.
  The patients will be placed on a table in ventral decubitus and the ankle outside the plane of the table in neutral position. To determine the point to be scanned, the maximum perpendicular distance between the anterior and posterior limits of the tendon between 2 to 6 cm from the insertion in the calcaneus will be taken and this value will be reported in mm.
  The SWS value will be expressed in m/s. The range of SWS is 0-9 m/s. The standard SWS measurement window size shall be 1cm2 , with a region of interest of 3mm. Three measurements will be recorded in each plane (regions of interest) where homogeneous tissue is considered and the average value of the 6 measurements will be reported.
ultrasound Shear Wave elastography - Week 8 | eight week at study entry
  Shear Wave Elastography (SWS), which consists of a special ultrasound methodology that allows quantitative characterization of the elastic capacity of a tissue through the propagation velocity of the ultrasound wave. The Siemens Acuson S2000 system with a model 9L4 linear transducer will be used.
  The patients will be placed on a table in ventral decubitus and the ankle outside the plane of the table in neutral position. To determine the point to be scanned, the maximum perpendicular distance between the anterior and posterior limits of the tendon between 2 to 6 cm from the insertion in the calcaneus will be taken and this value will be reported in mm.
  The SWS value will be expressed in m/s. The range of SWS is 0-9 m/s. The standard SWS measurement window size shall be 1cm2 , with a region of interest of 3mm. Three measurements will be recorded in each plane (regions of interest) where homogeneous tissue is considered and the average value of the 6 measurements will be reported.
ultrasound Shear Wave elastography - Week 12 | twelve week at study entry
  Shear Wave Elastography (SWS), which consists of a special ultrasound methodology that allows quantitative characterization of the elastic capacity of a tissue through the propagation velocity of the ultrasound wave. The Siemens Acuson S2000 system with a model 9L4 linear transducer will be used.
  The patients will be placed on a table in ventral decubitus and the ankle outside the plane of the table in neutral position. To determine the point to be scanned, the maximum perpendicular distance between the anterior and posterior limits of the tendon between 2 to 6 cm from the insertion in the calcaneus will be taken and this value will be reported in mm.
  The SWS value will be expressed in m/s. The range of SWS is 0-9 m/s. The standard SWS measurement window size shall be 1cm2 , with a region of interest of 3mm. Three measurements will be recorded in each plane (regions of interest) where homogeneous tissue is considered and the average value of the 6 measurements will be reported.
ultrasound Shear Wave elastography - Week 26 | twenty-six week at study entry
  Shear Wave Elastography (SWS), which consists of a special ultrasound methodology that allows quantitative characterization of the elastic capacity of a tissue through the propagation velocity of the ultrasound wave. The Siemens Acuson S2000 system with a model 9L4 linear transducer will be used.
  The patients will be placed on a table in ventral decubitus and the ankle outside the plane of the table in neutral position. To determine the point to be scanned, the maximum perpendicular distance between the anterior and posterior limits of the tendon between 2 to 6 cm from the insertion in the calcaneus will be taken and this value will be reported in mm.
  The SWS value will be expressed in m/s. The range of SWS is 0-9 m/s. The standard SWS measurement window size shall be 1cm2 , with a region of interest of 3mm. Three measurements will be recorded in each plane (regions of interest) where homogeneous tissue is considered and the average value of the 6 measurements will be reported.
ultrasound Shear Wave elastography - Week 52 | fifty-two week at study entry
  Shear Wave Elastography (SWS), which consists of a special ultrasound methodology that allows quantitative characterization of the elastic capacity of a tissue through the propagation velocity of the ultrasound wave. The Siemens Acuson S2000 system with a model 9L4 linear transducer will be used.
  The patients will be placed on a table in ventral decubitus and the ankle outside the plane of the table in neutral position. To determine the point to be scanned, the maximum perpendicular distance between the anterior and posterior limits of the tendon between 2 to 6 cm from the insertion in the calcaneus will be taken and this value will be reported in mm.
  The SWS value will be expressed in m/s. The range of SWS is 0-9 m/s. The standard SWS measurement window size shall be 1cm2 , with a region of interest of 3mm. Three measurements will be recorded in each plane (regions of interest) where homogeneous tissue is considered and the average value of the 6 measurements will be reported.
Vienna Achilles tendon morphological score - MRI - baseline | Baseline
  A 1.5T Siemens Healthcare 1.5T scanner will be used for the MRI evaluation, using a gradient strength of 40 mT/m and an 8-channel coil. The standard MRI protocol will be identical for all examinations and will consist of a localizer set and three morphological MR sequences: 1) a sagittal fat-suppressed sequence; 2) a sagittal T1 sagittal spin echo (SE) sequence and 3) a T2-w sequence.
  Once the images are obtained, they will be evaluated with the "Vienna Achilles tendon morphological score" (VIMATS) protocol proposed by Apprich S. (2021) which conforms a semiquantitative rating scale where the score is composed of four different parameters: (1) thickness, (2) continuity, (3) signal and (4) associated pathologies. It has a continuous numerical scale from 0 to 100 where the higher the score, the better the patient's stage.
Vienna Achilles tendon morphological score - MRI - Week 4 | four week at study entry
  A 1.5T Siemens Healthcare 1.5T scanner will be used for the MRI evaluation, using a gradient strength of 40 mT/m and an 8-channel coil. The standard MRI protocol will be identical for all examinations and will consist of a localizer set and three morphological MR sequences: 1) a sagittal fat-suppressed sequence; 2) a sagittal T1 sagittal spin echo (SE) sequence and 3) a T2-w sequence.
  Once the images are obtained, they will be evaluated with the "Vienna Achilles tendon morphological score" (VIMATS) protocol proposed by Apprich S. (2021) which conforms a semiquantitative rating scale where the score is composed of four different parameters: (1) thickness, (2) continuity, (3) signal and (4) associated pathologies. It has a continuous numerical scale from 0 to 100 where the higher the score, the better the patient's stage.
Vienna Achilles tendon morphological score - MRI - Week 8 | eight week at study entry
  A 1.5T Siemens Healthcare 1.5T scanner will be used for the MRI evaluation, using a gradient strength of 40 mT/m and an 8-channel coil. The standard MRI protocol will be identical for all examinations and will consist of a localizer set and three morphological MR sequences: 1) a sagittal fat-suppressed sequence; 2) a sagittal T1 sagittal spin echo (SE) sequence and 3) a T2-w sequence.
  Once the images are obtained, they will be evaluated with the "Vienna Achilles tendon morphological score" (VIMATS) protocol proposed by Apprich S. (2021) which conforms a semiquantitative rating scale where the score is composed of four different parameters: (1) thickness, (2) continuity, (3) signal and (4) associated pathologies. It has a continuous numerical scale from 0 to 100 where the higher the score, the better the patient's stage.
Vienna Achilles tendon morphological score - MRI - Week 12 | twelve week at study entry
  A 1.5T Siemens Healthcare 1.5T scanner will be used for the MRI evaluation, using a gradient strength of 40 mT/m and an 8-channel coil. The standard MRI protocol will be identical for all examinations and will consist of a localizer set and three morphological MR sequences: 1) a sagittal fat-suppressed sequence; 2) a sagittal T1 sagittal spin echo (SE) sequence and 3) a T2-w sequence.
  Once the images are obtained, they will be evaluated with the "Vienna Achilles tendon morphological score" (VIMATS) protocol proposed by Apprich S. (2021) which conforms a semiquantitative rating scale where the score is composed of four different parameters: (1) thickness, (2) continuity, (3) signal and (4) associated pathologies. It has a continuous numerical scale from 0 to 100 where the higher the score, the better the patient's stage.
Vienna Achilles tendon morphological score - MRI - Week 26 | twenty-six week at study entry
  A 1.5T Siemens Healthcare 1.5T scanner will be used for the MRI evaluation, using a gradient strength of 40 mT/m and an 8-channel coil. The standard MRI protocol will be identical for all examinations and will consist of a localizer set and three morphological MR sequences: 1) a sagittal fat-suppressed sequence; 2) a sagittal T1 sagittal spin echo (SE) sequence and 3) a T2-w sequence.
  Once the images are obtained, they will be evaluated with the "Vienna Achilles tendon morphological score" (VIMATS) protocol proposed by Apprich S. (2021) which conforms a semiquantitative rating scale where the score is composed of four different parameters: (1) thickness, (2) continuity, (3) signal and (4) associated pathologies. It has a continuous numerical scale from 0 to 100 where the higher the score, the better the patient's stage.
Vienna Achilles tendon morphological score - MRI - Week 52 | fifty-two week at study entry
  A 1.5T Siemens Healthcare 1.5T scanner will be used for the MRI evaluation, using a gradient strength of 40 mT/m and an 8-channel coil. The standard MRI protocol will be identical for all examinations and will consist of a localizer set and three morphological MR sequences: 1) a sagittal fat-suppressed sequence; 2) a sagittal T1 sagittal spin echo (SE) sequence and 3) a T2-w sequence.
  Once the images are obtained, they will be evaluated with the "Vienna Achilles tendon morphological score" (VIMATS) protocol proposed by Apprich S. (2021) which conforms a semiquantitative rating scale where the score is composed of four different parameters: (1) thickness, (2) continuity, (3) signal and (4) associated pathologies. It has a continuous numerical scale from 0 to 100 where the higher the score, the better the patient's stage.

CONTACTS AND LOCATIONS:
Overall Officials: Santiago M d'Almeida, PT SCS, Principal Investigator — Maimonides University
Locations (1):
- Maimonides University, Buenos Aires, Buenos Aires F.D., Argentina